CLINICAL TRIAL: NCT01189760
Title: Safety and Efficacy Study of Botulinum Toxin Type A for the Treatment of Crow's Feet Lines and Frown Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-099
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Facial Rhytides; Crow's Feet Lines; Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- onabotulinumtoxinA 44U (Experimental): 44 units (U) onabotulinumtoxinA (botulinum toxin Type A) total dose injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients received two treatments 4 months apart.
  Interventions: Biological: onabotulinumtoxinA 44 U
- onabotulinumtoxinA 24U (Other): 24 units onabotulinumtoxinA (botulinum toxin Type A) total dose and placebo (normal saline) injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients received two treatments 4 months apart.
  Interventions: Biological: onabotulinumtoxinA 24 U; Drug: normal saline
- placebo (normal saline) (Placebo Comparator): Normal Saline injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients received two treatments 4 months apart.
  Interventions: Drug: normal saline

INTERVENTIONS:
Biological: onabotulinumtoxinA 24 U — 24 units onabotulinumtoxinA (botulinum toxin Type A) total dose injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients will receive two treatments 4 months apart.
  Other Names: BOTOX®; BOTOX® Cosmetic; onabotulinumtoxinA
  Arms: onabotulinumtoxinA 24U
Biological: onabotulinumtoxinA 44 U — 44 units onabotulinumtoxinA (botulinum toxin Type A) total dose injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients will receive two treatments 4 months apart
  Other Names: BOTOX®; BOTOX® Cosmetic; onabotulinumtoxinA
  Arms: onabotulinumtoxinA 44U
Drug: normal saline — Normal Saline injected into bilateral Crow's Feet Line and Frown Line areas per treatment. Patients will receive two treatments 4 months apart.
  Arms: onabotulinumtoxinA 24U; placebo (normal saline)

SUMMARY:
This study will evaluate the safety and efficacy of botulinum toxin Type A compared to placebo for the treatment of Crow's Feet Lines and Frown Lines (Facial Rhytides)

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe Crow's Feet Lines and Frown Lines
* Have adequate vision without the use of eyeglasses to assess facial wrinkles in the mirror (contact lenses OK)

Exclusion Criteria:

* Current or previous botulinum toxin treatment of any serotype
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis
* Prior facial cosmetic surgery (e.g., prior periorbital surgery, facial lift, brow lift, eyelid lift or eyebrow surgery)
* Facial laser or light treatment, microdermabrasion, or superficial peels within 3 months
* Oral retinoid therapy within one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 917 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2011-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (4):
- Newport Beach, California, United States
- Vancouver, British Columbia, Canada
- Antibes, France
- Berlin, Germany

REFERENCES:
- [Background] Moers-Carpi M, Carruthers J, Fagien S, Lupo M, Delmar H, Jones D, Somogyi C, Lee E, Lei X, MacKinnon S, Davis PG, Yalamanchili R, Campo A, Beddingfield FC 3rd. Efficacy and safety of onabotulinumtoxinA for treating crow's feet lines alone or in combination with glabellar lines: a multicenter, randomized, controlled trial. Dermatol Surg. 2015 Jan;41(1):102-12. doi: 10.1097/DSS.0000000000000220. PMID 25485803

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline)
Started | 305 | 306 | 306
Completed | 291 | 283 | 255
Not Completed | 14 | 23 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 305 | 306 | 306 | 917
Age, Customized [Number; unit: Participants]
  <45 Years | 87 | 89 | 100 | 276
  45 to 65 Years | 204 | 200 | 194 | 598
  >65 Years | 14 | 17 | 12 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 267 | 273 | 263 | 803
  Male | 38 | 33 | 43 | 114
CFL Severity as Assessed by the Investigator [Number; unit: Participants] — Crow's Feet Line (CFL) severity as assessed at Baseline by the Investigator using the 4-point Facial Wrinkle Scale (FWS) at maximum smile.
  Participants
    Moderate | 109 | 115 | 113 | 337
    Severe | 196 | 191 | 193 | 580

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders Based on Composite Facial Wrinkle Scale Assessment of Crow's Feet Line Severity at Maximum Smile
Description: The composite facial wrinkle scale assessment is based on both the Investigator and Subject Facial Wrinkle scales at Day 30. The Investigator assessed the severity of the patient's Crow's Feet Lines at maximum smile using the 4-point Facial Wrinkle Scale: 0=none, 1=mild, 2=moderate or 3=severe and the patient assessed the severity of their Crow's Feet Lines at maximum smile using the same 4-point Facial Wrinkle Scale. A responder is defined as a participant with a ≥ 2-grade improvement from Baseline.
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all randomized participants. Participants with missing values are considered non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline)
Number analyzed (Participants) | 305 | 306 | 306
Percentage of participants | 21.3 | 20.6 | 0.0

2. Secondary Outcome: Percentage of Participants Achieving a Grade of None or Mild at Maximum Smile Based on the Investigator Facial Wrinkle Scale Assessment of the Severity of Crow's Feet Lines
Description: The Investigator assessed the severity of the patient's Crow's Feet lines at maximum smile using the 4-point Facial Wrinkle Scale: 0=none, 1=mild, 2=moderate or 3=severe. The percentage of participants with a score of none or mild at Day 30 is reported.
Time Frame: Day 30
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline)
Number analyzed (Participants) | 305 | 306 | 306
Percentage of participants | 59.0 | 54.9 | 3.3

3. Secondary Outcome: Percentage of Participants With a ≥ 1-Grade Improvement From Baseline by Investigator Facial Wrinkle Scale Assessment of the Severity of Crow's Feet Lines at Maximum Smile
Description: The Investigator assessed the severity of the patient's Crow's Feet Lines at maximum smile using the 4-point Facial Wrinkle Scale: 0=none, 1=mild, 2=moderate or 3=severe. The percentage of participants with a ≥ 1-grade improvement from Baseline at Day 30 is reported.
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline)
Number analyzed (Participants) | 305 | 306 | 306
Percentage of participants | 87.9 | 78.1 | 10.1

4. Secondary Outcome: Percentage of Participants With a ≥ 1-Grade Improvement From Baseline by Investigator Facial Wrinkle Scale Assessment of the Severity of Crow's Feet Lines at Rest
Description: The Investigator assessed the severity of the patient's Crow's Feet Lines at rest using the 4-point Facial Wrinkle Scale: 0=none, 1=mild, 2=moderate or 3=severe. The percentage of participants with a ≥ 1-grade improvement from Baseline at Day 30 is reported.
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all randomized participants. Only those participants who were rated at least mild at Baseline are included in the analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline)
Number analyzed (Participants) | 293 | 297 | 298
Percentage of participants | 75.1 | 61.3 | 13.4

5. Secondary Outcome: Subject Global Assessment of Change in Crow's Feet Lines (SGA-CFL) Score
Description: Patients rated the change in their Crow's Feet Lines using the SGA-CFL 7-point scale: 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse or 7=very much worse at Day 30. Lower scores indicate improvement.
Time Frame: Day 30
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline)
Number analyzed (Participants) | 305 | 306 | 306
Score on a scale | 2.3 (0.96) | 2.5 (1.05) | 3.8 (0.54)

6. Secondary Outcome: Percentage of Participants Who Judged Themselves in a Younger Self-Perception of Age Category Than at Baseline
Description: Participants were considered to judge themselves as looking younger if the category change was from "look my current age" at Baseline to "look younger" at Day 30 or from "look older" at Baseline to "look my current age/younger" at Day 30.
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all randomized participants. Only those participants who rated themselves as "look my current age" or "look older" at Baseline are included in the analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline)
Number analyzed (Participants) | 265 | 265 | 263
Percentage of participants | 50.6 | 33.6 | 9.1

7. Secondary Outcome: Percentage of Participants With a ≥ 2-point Improvement From Baseline for Facial Line Outcomes Questionnaire (FLO-11) Item 2 at Day 30
Description: The percentage of FLO-11 Item #2 responders, defined as participants with a ≥ 2-point improvement in FLO-11 score from Baseline for FLO-11 Question #2: "When I look in the mirror, my facial lines make me look older than I want to look." The FLO-11 questionnaire is comprised of 11 items that assess the subject's perceptions about specific aspects of their facial lines for the previous 7 days. Each question is scored on an 11-point scale (0=not at all, 5=somewhat, 10=very much).
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all randomized participants. Only participants with a Baseline score ≥ 2 are included.
Measure: Number; unit: Percentage of participants
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline)
Number analyzed (Participants) | 292 | 298 | 293
Percentage of participants | 69.9 | 54.4 | 24.6

8. Secondary Outcome: Percentage of Participants With a ≥ 2-point Improvement From Baseline for Facial Line Outcomes Questionnaire (FLO-11) Item 5 at Day 30
Description: The percentage of FLO-11 Item #5 responders, defined as participants with a ≥ 2-point improvement in FLO-11 score from Baseline for FLO-11 Question #5: "My facial lines make me look less attractive than I want to look." The FLO-11 questionnaire is comprised of 11 items that assess the subject's perceptions about specific aspects of their facial lines for the previous 7 days. Each question is scored on an 11-point scale (0=not at all, 5=somewhat, 10=very much).
Time Frame: Baseline, Day 30
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline)
Number analyzed (Participants) | 287 | 282 | 280
Percentage of participants | 61.7 | 48.6 | 18.6

9. Secondary Outcome: Percentage of Participants With a ≥ 3-point Improvement From Baseline for Facial Line Outcomes Questionnaire (FLO-11) Item 8 at Day 30
Description: The percentage of FLO-11 Item #8 responders, defined as participants with a ≥ 3-point improvement in FLO-11 score from Baseline for FLO-11 Question #8: "My facial lines make me look tired." The FLO-11 questionnaire is comprised of 11 items that assess the subject's perceptions about specific aspects of their facial lines for the previous 7 days. Each question is scored on an 11-point scale (0=not at all, 5=somewhat, 10=very much).
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all randomized participants. Only participants with a Baseline score ≥ 3 are included.
Measure: Number; unit: Percentage of participants
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline)
Number analyzed (Participants) | 284 | 280 | 282
Percentage of participants | 58.1 | 40.7 | 14.9

ADVERSE EVENTS:
Description: The safety population (all randomized and treated participants) was used to calculate the number of participants at risk for Serious Adverse Events and Adverse Events.
Arm/Group | onabotulinumtoxinA 44U | onabotulinumtoxinA 24U | Placebo (Normal Saline)
Serious Adverse Events (participants affected / at risk) | 5/305 | 8/306 | 6/306
Other Adverse Events (participants affected / at risk) | 58/305 | 51/306 | 38/306
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | onabotulinumtoxinA 44U (N=305) | onabotulinumtoxinA 24U (N=306) | Placebo (Normal Saline) (N=306)
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Goitre (Endocrine disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Breast cellulitis (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | onabotulinumtoxinA 44U (N=305) | onabotulinumtoxinA 24U (N=306) | Placebo (Normal Saline) (N=306)
Nasopharyngitis (Infections and infestations) | 24 | 18 | 15
Headache (Nervous system disorders) | 19 | 14 | 18
Injection site haematoma (General disorders) | 15 | 19 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.